CLINICAL TRIAL: NCT04551612
Title: Evaluation of the Level of Middle Cranial Fossa Dura in Patients With Cholesteatoma
Brief Title: Level of Middle Cranial Fossa Dura in Patients With Cholesteatoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Zakaria, Principal investigator, Assiut University
Other Study IDs: Patients with Cholesteatoma
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Cholesteatoma, Middle Ear
MeSH Terms: conditions — Cholesteatoma, Middle Ear

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cholesteatoma: Patients with cholesteatoma in one ear that will compared with the other healthy one.
  Interventions: Radiation: Multislice computed tomography temporal bone

INTERVENTIONS:
Radiation: Multislice computed tomography temporal bone — Patients with cholesteatoma will undergo multislice computed tomography (MSCT) temporal bone images. Then The Tegmen level will be determined and compared with the other normal ear at the same patient

SUMMARY:
Cholesteatoma is a destructive lesion that progressively expands in the middle ear, mastoid or petrous bone and leads to destruction of the nearby structures. Erosion, which is caused by bone resorption of the ossicular chain and otic capsule, may cause hearing loss, vestibular dysfunction, facial paralysis and intracranial manifestations

DETAILED DESCRIPTION:
Cholesteatoma has three Classical forms: (1) Congenital, primary or genuine cholesteatoma: occurs behind an intact tympanic membrane. Primary acquired cholesteatoma: looks like a limited diverticulum of the pars flaccida with little or no history of otorrhea. Secondary acquired cholesteatoma: develops with posterosuperior perforations in eardrum and expansion of the disease process into the antrum, mastoid, attic and middle ear. Granulation tissue, polyps and foul- smelling otorrhea are common findings in this type

ELIGIBILITY:
Inclusion Criteria:

* All adults above the age of 18 presented to the Assiut university Clinic with

cholesteatoma will be included in the study.

Exclusion Criteria:

1. Patients with previous mastoid surgery
2. Patients with Craniofacial anomalies or cleft lip and palate
3. Pediatric populations ≤ 18 years old
4. Patients with congenital ear anomalies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cholesteatoma in one ear
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Level of Middle Cranial Fossa Dura in Patients with Cholesteatoma by multislice computed tomography. | One year
  determination the level of tegmen in patients with attico-antral diseases by MSCT